CLINICAL TRIAL: NCT03977766
Title: Feasibility of a Process of Digital Validation of Outpatients Chemotherapies in a Day Treatment Unit
Brief Title: Feasibility of a Process of Digital Validation of Chemotherapies in a Day Treatment Unit
Acronym: CPV2-0
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CPV 2.0-IPC 2018-054
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Solid Tumor, Adult
Keywords: digital application; outpatients chemotherapy; chemotherapy validation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nurse then patient digital prevalidation of chemotherapy (Experimental): Outpatient Chemotherapy prevalidation will done
  * with the help of a nurse, using the digital application, for cycle 2 and 3.
  * by the patient alone, using the digital application, for cycle 4 and 5.
  Interventions: Procedure: Chemotherapy prevalidation

INTERVENTIONS:
Procedure: Chemotherapy prevalidation — Outpatient Chemotherapy prevalidation will done
  * with the help of a nurse, using the digital application, for cycle 2 and 3.
  * by the patient alone, using the digital application, for cycle 4 and 5.

SUMMARY:
The aim of CPV 2.0 study is to evaluate a process of digital prevalidation of outpatients chemotherapy thanks to a numeric application. This digital tool is based on the combination of the US National Cancer Institute's Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) to a decisional algorithm.

After cycle 1, chemotherapy digital prevalidation will be done with the help of a nurse for two consecutive cycles (cycles 2 and 3). Patients will then have to use to application by themselves for the two following cycles (cycles 4 and 5)

ELIGIBILITY:
Inclusion Criteria:

* Age <80 (if age>70 years, a G8 score>14 is required)
* ECOG<3
* Pathology (solid tumor, in neoadjuvant, adjuvant or metastatic setting)
* Patient receiving an IV cytotoxic chemotherapy in a day treatlent unit for at least 5 cycles, with at least an injection at day 1, day 8 and day 15
* Familiar with digital tools

Exclusion Criteria:

* Emergency
* patient feeling unease with the use of a smartphone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2021-04-15 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the digital application | 6 weeks
  Number of prevalidation of the chemotherapy by the digital application compared to the number of corresponding validation of the chemotherapy by the physician

CONTACTS AND LOCATIONS:
Overall Officials: Loui Tassy, Principal Investigator — Institut Paoli-Calmettes